CLINICAL TRIAL: NCT06239129
Title: The Stockholm CREAtinine Measurements (SCREAM) Project
Brief Title: The Stockholm CREAtinine Measurements Project
Acronym: SCREAM
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Juan Jesus Carrero, Professor of Cardiorenal Epidemiology, Karolinska Institutet
Other Study IDs: 000001
Record Dates: First submitted 2024-01-17; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Chronic Kidney Diseases; Acute Kidney Injury; Diabetes Mellitus; Cardiovascular Diseases; Hypertension
MeSH Terms: conditions — Renal Insufficiency, Chronic; Acute Kidney Injury; Diabetes Mellitus; Cardiovascular Diseases; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Initiation of specific medications — multiple therapies studied within this database
  Other Names: multiple therapies studied within this database
Procedure: Undertaking of specific procedures — multiple procedures/surgeries studied within this database
Diagnostic Test: Abnormalities in specific laboratory tests — multiple abnormalities in laboratory values (i.e. CRP, cholesterol, eGFR, potassium) studied within this database

SUMMARY:
The Stockholm CREAtinine Measurements (SCREAM) project is a healthcare utilization cohort including, at present, all adult residents in Stockholm between 2006 and 2021. The region of Stockholm had a population of 2.3 million citizens in 2021and provides universal healthcare with a single unified health-system. Administrative databases with complete information on socidemographic data, healthcare use, diagnoses and therapeutic/surgical procedures, and vital status were enriched with performed laboratory tests, dispensed prescriptions at Swedish pharmacies and validated kidney replacement therapy endpoints. Registries were linked and de-identified by the Swedish National Board of Welfare and are considered to have no or minimal loss to follow-up. Because the study utilized de-identified data, it was deemed not to require informed consent and was approved by the regional ethical review boards and the Swedish National Board of Welfare.

For detailed description of available data and linked registers please consult:

https://pubmed.ncbi.nlm.nih.gov/35028991/

DETAILED DESCRIPTION:
Please consult cohort description in:

https://pubmed.ncbi.nlm.nih.gov/35028991/ https://pubmed.ncbi.nlm.nih.gov/26798472/

ELIGIBILITY:
Inclusion Criteria:

For both cohorts:

Be a resident of Stockholm during 2006-2021, of all ages

For the primary cohort:

To have undertaken at least one test of serum creatinine or albuminuria during 2006-2021. If this condition is met, we will then extract a broad range of laboratory tests

For the secondary cohort:

Anyone not undertaking a test of serum creatinine or albuminuria will conform the secondary cohort. In this cohort we will not extract any other laboratory test, but will obtain the rest of healthcare information

Exclusion criteria:

None

Ages: 0 Years to 110 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Stockholm residents with/without ever testing for creatinine or albumuninuria
Sampling Method: Non-Probability Sample
Enrollment: 3200000 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Adverse health events by levels of kidney function | 2006-2021
  multiple outcomes evaluated such as cardiovascular events, fractures, dementia, cancer, etc, all of them based on claims data and/or laboratory data
Safety and efficacy of medications by levels of kidney function | 2006-2021
  multiple outcomes evaluated depending on the treatments of interest, all of them based on claims data and/or laboratory data
Effect of medications or conditions on kidney function decline | 2006-2021
  Evaluation of changes in kidney function over time upon occurrence of a certain condition (i.e., heart failure or covid19 infection) or initiation of a specific medication

SECONDARY OUTCOMES:
Adverse health events associated to laboratory abnormalities | 2006-2021
  Same as primary objectives but for other laboratory abnormalities different from kidney function measures

CONTACTS AND LOCATIONS:
Overall Officials: Juan J Carrero, Prof, Principal Investigator — Karolinska Institutet

IPD SHARING:
Plan to Share IPD: Yes
Possibility to share data for collaborative academic research purposes that comply with institutional, national and international ethic principles and legislation on data sharing, access and investigation
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: For the time required to perform the collaborative project
Access Criteria: Primarily by welcoming researchers to analyse the data physically in Stockholm. Exceptionally by opening secure VDI connections to work under our online servers

REFERENCES:
- [Derived] Russel WA, Fu EL, Bosi A, Caldinelli A, Inker LA, Chang AR, Levey AS, Carrero JJ. Obesity, Underweight, and Accuracy of eGFR Using Cystatin C and Creatinine in a Northern European Population. J Am Soc Nephrol. 2025 Nov 1;36(11):2177-2189. doi: 10.1681/ASN.0000000760. Epub 2025 Jun 13. PMID 40512561